CLINICAL TRIAL: NCT04793087
Title: Post-COntrast 3D SE T1 Versus Coronal SE T1-WI MRI in Detecting Optic Neuritis in Patients Presenting With Acute Visual Loss and Otherwise Normal Ophthalmological Examination
Brief Title: Post-COntrast 3D SE T1 Versus Coronal SE T1-WI MRI in Detecting Optic Neuritis (COCON)
Acronym: COCON
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20200204_2_ALR
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Optic Neuritis; Multiple Sclerosis
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Comparing 3D T1 versus coronal T1 MRI in detecting Optic Neuritis

SUMMARY:
3D FLAIR, 3D T1 FAT SAT, coronal T2 and coronal T1 dixon sequences were usually used to assess visual deficits in MRI. Optic nerve examination is preferably performed using a coronal T2 sequence in order to detect a hypersignal suggestive of inflammation whereas brain examination is preferably performed using a 3D T1 sequence to highlight signs of spatial dissemination and lesions suggestive of multiple slerosis (MS). No study has yet investigated the detection capabilities of 3D T1 for the detection of optic nerve inflammation. The objective of this retrospective study was to determine whether a single 3D T1 sequence allows simultaneous exploration of the optic nerve and the brain for the positive diagnosis of optic neuropathy and/or MS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Decrease in visual acuity explored in MRI between january 2018 and january 2020

Exclusion Criteria:

* Past history of episode of Optic neuritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with visual acuity loss explored by MRI between january 2018 and january 2020
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Detection of optic neuropathies using MRI | 1 hour
  MRI comparison of the diagnostic performance of the 3D T1 sequence and the T1 coronal in the detection of optic neuropathies.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France